CLINICAL TRIAL: NCT07061639
Title: A Phase 1/2 Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of QLS5133 Monotherapy in Subjects With Advanced Solid Tumors
Brief Title: A Study of QLS5133 Monotherapy in Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: QLS5133-101
Record Dates: First submitted 2025-07-01; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Monotherapy Dose Finding (Experimental)
  Interventions: Drug: QLS5133
- PK expansion as Monotherapy (Experimental)
  Interventions: Drug: QLS5133
- Cohort expansion as Monotherapy (Experimental)
  Interventions: Drug: QLS5133

INTERVENTIONS:
Drug: QLS5133 — antibody drug conjugate (ADC)

SUMMARY:
The phase 1/2 clinical study includes three stages: Phase 1 dose escalation, phase 1 PK expansion and phase 2 cohort expansion：

* Phase 1: Assesse safety, tolerability, PK, immunogenicity and preliminary efficacy of QLS5133 in advanced solid tumors. Phase 1 dose escalation will use ATD + BOIN, the maximum sample size for each dose group is 12. For Phase 1 PK expansion, 1 to 4 appropriate doses will be selected. After the DLT observation period in the selected dose group up to 12 subjects (including those subjects in the dose escalation stage) can be further enrolled for PK expansion.
* Phase 2: Evaluates QLS5133's anti-tumor efficacy in subjects with advanced solid tumors. at least 2 dose groups will be expanded.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥ 18 years on the day of signing the ICF, male or female;
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) score: 0 or 1;
* Measurable disease, per RECIST v1.1;
* Adequate organ function;
* Recover from all reversible AEs from previous anti-tumor treatment (i.e., Grade ≤ 1, according to NCI-CTCAE v5.0), excluding alopecia (any grade) and Grade ≤ 2 neuropathy peripheral, or who experience other abnormalities that are not clinically significant or toxicities judged to have no risk by the investigator;
* Left ventricular ejection fraction (LVEF) ≥ 50%;

Exclusion Criteria:

* Previous treatment with drugs targeting CDH6 (including ADCs), or any drug containing topoisomerase I inhibitors (including ADCs);
* Large and uncontrollable pleural, pericardial or abdominal effusion before the first dose (those who are stable for at least 2 weeks after drainage can be enrolled);
* Progressive or symptomatic brain metastases;
* Clinically significant bleeding symptoms or obvious bleeding tendency within 1 month before the first dose
* History of significant cardiac disease, or poorly controlled diabetes mellitus;
* History of recurrent autoimmune diseases;
* History of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML);
* History of other active malignant tumors within 3 years before signing the informed consent form;
* If female, is pregnant or breastfeeding;
* Be allergic to any component of QLS5133 or its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Estimated)
Dates: Start 2025-07 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and serious adverse events | up to 2 years
  Incidence and severity of adverse events, serious adverse events, according to NCI-CTCAE Version 5.0
Maximum tolerated dose (MTD) | 28days
  Highest administered dose with < 33% participants experiencing dose limiting toxicity (DLT) in the first 6 DLT evaluable participants
Recommended Phase 2 Dose (RP2D) | up to 2 years
  Based on the maximum tolerated dose, cumulative safety, and pharmacokinetic data
Objective Response Rate (ORR) | up to 2 years
  Percentage of participants with best response of complete response (CR) or partial response (PR) according to RECIST 1.1

SECONDARY OUTCOMES:
Maximum Serum Concentration of QLS5133 (Cmax) | 21 days
  PK assessment
Maximum Serum Concentration of QLS5133 at Steady State (Cmax,ss) | 63 days
  PK assessment
Minimum Serum Concentration of QLS5133 at Steady State (Cmin,ss) | 63 days
  PK assessment
Time of Maximum Serum Concentration of QLS5133 (Tmax) | 21 days
  PK assessment
Terminal Half-life (T1/2) of Serum QLS5133 | 63 days
  PK assessment
Area under the Serum Concentration-Time curve from the time of dosing to the last measurable concentration (AUC0-t) for QLS5133 | 21 days
  PK assessment
Area under the Serum Concentration-Time curve from the time of dosing extrapolated to time infinity (AUC0-∞) for QLS5133 | 63 days
  PK assessment
Apparent Volume of Distribution (Vd) of QLS5133 | 63 days
  PK assessment
Clearance (CL) of QLS5133 | 63 days
  PK assessment
Duration of Response (DOR) | up to 2 years
  Time from CR or PR to objective disease progression or death to any cause
Progression Free Survival (PFS) | up to 2 years
  PFS is defined as the time from the start of the treatment until objective disease progression or death from any cause
Time to Progression (TTP) | 1 years
  Time from start of treatment to disease progression
1 Year Overall Survival (1YOS) | 1 years
  Proportion of participants alive at 1 year from the start of treatment to death from any cause
2 Year Overall Survival (2YOS) | 2 years
  Proportion of participants alive at 2 years from the start of treatment to death from any cause
Number of anti-drug antibody (ADA) Positive Participants | up to 2 years
  Immunogenicity will be measured by the number of participants that are ADA positive
Number of neutralizing antibody (Nab) Positive Participants | up to 2 years
  Immunogenicity will be measured by the number of participants that are Nab positive

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China